CLINICAL TRIAL: NCT06662227
Title: A Clinical Study Evaluating the Safety and Efficacy of Universal CD19-Targeted CAR-T (UWD-CD19) Therapy for Refractory and Relapsed B-Cell Tumors
Brief Title: Universal CAR-T Cells (REVO-UWD-19) for Refractory and Relapsed B-Cell Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wondercel Biotech (ShenZhen) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-REVO-UWD-19
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: B Cell Lymphoma; B Cell Leukemia; B Cell Malignancy
Keywords: CAR-T; Universal CAR-T; CD19; B cell lymphoma; B cell leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Off-the-shelf REVO-UWD-19 (Experimental): Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning, followed by a one-time injection of universal UWD-19 cells
  Interventions: Biological: Single dose injection of certain dose of UWD-19; Drug: MMF Immunosuppression

INTERVENTIONS:
Biological: Single dose injection of certain dose of UWD-19 — Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning after signing an informed consent form, followed by a one-time injection of certain dose of universal UWD-19 cells
Drug: MMF Immunosuppression — One day after the completion of fludarabine preconditioning (D-2), initiate oral mycophenolate sodium at a dose of 1440 mg twice daily (BID) for 15 consecutive days, or extend the duration appropriately based on CAR-T cell expansion status (discontinuation may occur at the end of CAR-T cell expansion or on the day of patient discharge). The maximum duration of administration must not exceed 30 days.

SUMMARY:
This study is a single-arm, single-center, investigator-initiated clinical trial. The primary objective is to evaluate the safety and preliminary efficacy of administering universal CD19 CAR-T cells to subjects with refractory and relapsed B-cell tumors. Eligible participants will undergo FC lymphodepleting chemotherapy preconditioning after signing an informed consent form, followed by a one-time injection of universal UWD-19 to assess its safety and efficacy. Subjects will be hospitalized for a period, and after discharge, they will undergo periodic efficacy assessments and long-term survival follow-up for at least five years.

DETAILED DESCRIPTION:
This study is a single-arm clinical trial evaluating the universal CD19-targeted CAR-T cell therapy (UWD-CD19) in treating relapsed and refractory B-cell tumors. Initiated by investigators, the study aims to assess the safety and preliminary efficacy of this cell therapy, providing new therapeutic options for patients with B-cell tumors-a class of hematologic malignancies that often recur and resist standard treatments, posing substantial treatment challenges.

CD19 is a specific marker predominantly expressed on the surface of B-cells, making it a prime target for CAR-T cell therapies. CAR-T therapy involves extracting T cells from a healthy donor and genetically engineering them to recognize and attack CD19-expressing tumor cells. UWD-CD19, a "universal" CAR-T cell product, seeks to enhance therapy adaptability, allowing it to effectively target B-cell tumors across different patient groups.

Study Objectives The primary objective of this study is to observe the therapeutic response in patients with relapsed or refractory B-cell tumors through a single infusion of UWD-CD19, specifically focusing on safety, tolerability, and preliminary efficacy. The research team will also conduct long-term follow-up on patients to assess the durability of treatment effects and survival rates, providing data support for the potential wider application of this novel therapy.

Inclusion Criteria: Patients aged between 3 and 70, with no gender restrictions, must meet diagnostic criteria for B-cell lymphoma with CD19-positive tumor cells. Patients should have an evaluable or measurable lesion as defined by the 2014 Lugano criteria.

Preconditioning: Eligible patients will receive lymphodepleting chemotherapy with Fludarabine and Cyclophosphamide before cell infusion to suppress the immune system and optimize CAR-T cell performance.

CAR-T Cell Infusion: Patients will receive a one-time infusion of UWD-CD19 cells, and their responses will be closely monitored during and after infusion to ensure safety.

Follow-up and Efficacy Assessment: Following treatment, patients will be hospitalized for a period and, after discharge, return regularly for follow-up and efficacy evaluations. The research team will conduct survival monitoring for at least five years.

Inclusion and Exclusion Criteria To ensure the study's safety and scientific rigor, strict inclusion and exclusion criteria are set. Patients must meet requirements across age, pathology, disease stage, and organ function, and should not have other severe health conditions (e.g., active CNS involvement, severe cardiovascular disease, serious infections) that could confound efficacy assessments or increase patient risk.

Potential Impact If results demonstrate good safety and efficacy of UWD-CD19 cell therapy in patients with relapsed and refractory B-cell tumors, this could open a new treatment pathway for this patient population. Universal CAR-T cell therapy could eventually extend to more hematologic malignancies, offering hope and support to patients facing significant treatment barriers.

Ethics and Risk Management The study has been approved by the Medical Ethics Committee, and the research team will strictly adhere to ethical standards, ensuring patients provide informed consent and receive adequate medical support. Since CAR-T therapy may present potential side effects (e.g., cytokine release syndrome, neurotoxicity), patients will be under real-time monitoring, with prompt intervention provided as needed.

This study aims to provide new insights and therapeutic approaches for B-cell tumor treatment through an in-depth evaluation of UWD-CD19 cell therapy. The research team will continue observing and recording patients' responses, establishing a scientific foundation for future immunotherapies in oncology and offering patients the prospect of long-term health benefits and quality of life improvements.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or their guardians) understand the study and voluntarily sign the informed consent form, with an expected ability to complete follow-up evaluations and treatments as per study protocol.

Age range: 3-70 years, no gender restrictions. Diagnosis of B-cell lymphoma, meeting the 2018 NCCN B-Cell Lymphoma guidelines (Version 5), with CD19 positivity confirmed by flow cytometry or immunohistochemistry.

At least one evaluable or measurable lesion per Lugano 2014 criteria. Evaluable lesions are indicated by FDG uptake above liver levels on FDG/PET or by lymphoma-like characteristics on PET/CT. Measurable lesions require a nodal diameter >15 mm or extranodal lesion >10 mm (with post-radiation evidence of progression if previously irradiated). Cases without measurable lesions but with diffuse liver FDG uptake are excluded.

Refractory and relapsed B-cell lymphoma, meeting at least one of the following: a. Received ≥2 cycles of standardized second-line or higher treatment, and meets Lugano 2014 criteria for best clinical response:

Progressive Disease (PD) on the most recent treatment.

Stable Disease (SD) lasting <6 months before progressing. b. Recurrence or progression ≤12 months post-autologous stem cell transplant. c. Based on investigator judgment, the potential benefit may outweigh risk in cases such as:

Recent SD with measurable disease progression but not meeting PD criteria. Partial remission (PR) or better lasting <6 months post-treatment, then progression.

Intolerance to most recent chemotherapy. Relapsed/refractory CD19-positive acute B lymphoblastic leukemia.

Laboratory values indicating adequate organ and marrow function, with no severe cardiac, pulmonary, hepatic, renal, or immune dysfunction:

Serum albumin ≥25 g/L Creatinine clearance ≥30 mL/min/1.73 m² ALT and AST ≤3.0× ULN Total bilirubin ≤2.0× ULN (exceptions for congenital hyperbilirubinemia like Gilbert syndrome with direct bilirubin ≤1.5× ULN) PT and APTT <2× ULN Oxygen saturation ≥95% Blood transfusions allowed to maintain hemoglobin ≥8.0 g/dL. ECOG performance status 0-1. Expected survival time >90 days. Negative β-hCG test for women of childbearing potential at screening and prior to chemotherapy.

Women of childbearing potential must use a highly effective contraceptive method (annual failure rate <1%) from the time of consent until 1 year after UWD-CD19 infusion, including:

Non-user-dependent: implantable progestogen, IUD, hormone-releasing system, or partner vasectomy.

User-dependent: combination hormonal contraception, progestogen-only pill, or injection.

Exclusion Criteria:

* History of aggressive malignancies other than B-cell lymphoma, except:

Cancer in remission >2 years post-curative therapy. Non-melanoma skin cancer successfully treated and inactive.

Prior anti-cancer therapy including:

Targeted, epigenetic, or experimental drug therapy within 14 days or 5 half-lives.

Cytotoxic therapy within 14 days. Immunomodulators within 7 days. Monoclonal antibodies within 21 days. Radiotherapy within 14 days. Active CNS involvement. Conditions like Waldenström's macroglobulinemia, POEMS syndrome, or primary AL amyloidosis.

Active hepatitis B (HBsAg or HBcAb positive with viral load >1000 copies/ml), hepatitis C (HCV RNA positive), HIV, CMV, or syphilis positivity.

Severe allergy history, or known allergy to trial components, adjuvants, or animal-derived proteins.

Severe cardiac conditions such as arrhythmias, unstable angina, recent MI, heart failure (NYHA III/IV), uncontrolled hypertension.

Unstable systemic disease, including significant liver, kidney, or metabolic disease requiring medication.

Acute/chronic GVHD or requiring immunosuppressants within 6 months. Active autoimmune or inflammatory neurologic diseases. Urgent tumor-related conditions requiring emergency treatment. Uncontrolled bacterial, fungal, or viral infections. Major surgery within 4 weeks or planned major surgery during the study. Live virus vaccination within 4 weeks prior to screening. Severe psychiatric disorders. History of substance abuse. Pregnant or lactating women, or individuals planning conception within 2 years of cell infusion.

Any contraindications per investigator's judgment due to clinical standards or patient's condition.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | [Time Frame: Within the first month post-infusion.]
  The highest dose of UWD-19 CAR-T cells that can be administered without causing unacceptable side effects, measured during the dose escalation phase.
Dose-Limiting Toxicities (DLT) | [Time Frame: Within the first month post-infusion.]
  The incidence of treatment-related toxicities that prevent further dose escalation.
Treatment-Emergent Adverse Events (TEAE) | [Time Frame: From the administration of UWD-19 CAR-T cells through six months post-infusion]
  The frequency and severity of adverse events that arise following the administration of UWD-19-CAR-T cells.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | [Time Frame: Measured at 3 and 6 months after treatment.]
  The proportion of patients with a measurable reduction in tumor size (complete or partial response) following UWD-19 CAR-T therapy.
Progression-Free Survival (PFS) | [Time Frame: From the start of treatment up to 5 years.]
  The length of time during and after treatment that the patient lives without disease progression.
Overall Survival (OS) | [Time Frame: From the start of treatment up to maximum follow-up period of five years.]
  The duration from the start of treatment to the time of death from any cause.
Duration of Response (DOR) | [Time Frame: From the administration of UWD-19 CAR-T cells to a maximum follow-up period of five years.]
  The time from initial tumor response (CR or PR) to disease progression or relapse or any cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, M.D. Ph.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No